CLINICAL TRIAL: NCT01495910
Title: An Open-Label, Multiple-Dose, Dose-Finding Study of Abiraterone Acetate in Adult Women With 21-Hydroxylase Deficiency
Brief Title: A Study Examining Doses of Abiraterone Acetate in Adult Women With 21-Hydroxylase Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100007; 212082HPL1002 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2011-11-23; First posted 2011-12-20 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: 21-hydroxylase Deficiency
Keywords: 21-hydroxylase deficiency; Androstenedione; Abiraterone acetate; Pharmacokinetics; Pharmacodynamics; Dose-finding
MeSH Terms: conditions — Congenital adrenal hyperplasia due to 21 hydroxylase deficiency | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abiraterone acetate (Experimental): Abiraterone acetate oral suspension administered daily from study Day 1 to study Day 6 of each treatment period: the first dose level is 100 mg with escalating doses of 250 mg and 500 mg in subsequent treatment periods.
  Interventions: Drug: Abiraterone acetate

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate oral suspension administered daily from study Day 1 to study Day 6 of each treatment period: the first dose level is 100 mg with escalating doses of 250 mg and 500 mg in subsequent treatment periods.

SUMMARY:
The purpose of this study is to determine the minimum dose of abiraterone acetate needed to decrease serum androstenedione to age-appropriate levels in premenopausal women on steroid replacement for classic 21-hydroxylase deficiency.

DETAILED DESCRIPTION:
This is a non-randomized (patients will not be assigned by chance to study treatments), open-label (patients will know the identity of study treatments), multiple-dose, intra-patient sequential dose-escalation study with a planned enrollment of approximately 10 patients. This study will consist of a screening period and a treatment period. Due to the intra-patient dose escalation, there will be multiple treatment periods consisting of 8 days each. A rest period of at least 7 days will separate each treatment period. Eligible patients will take study-defined replacement doses of hydrocortisone and fludrocortisone. Abiraterone acetate oral suspension will be administered in daily escalating doses from 100 mg to 500 mg. Patients will proceed to the next higher dose level when the majority of the treated patients have a reduction in the androstenedione level. Serial pharmacokinetic (study of what the body does to a drug) and pharmacodynamic (study of the effects of a drug on the body) samples will be collected at each treatment period as detailed in the protocol. All patients who receive at least 1 dose of abiraterone acetate will be analyzed for safety.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women >=18 years of age.
* Must be receiving a hormonal contraceptive agent containing both estrogen and progesterone.
* Confirmed 21-hydroxylase deficiency by CYP21A2 genotype associated with classic congenital adrenal hyperplasia.
* Demonstrates a >=1.5 X ULN of morning serum androstenedione concentration while taking study-defined doses of hydrocortisone and fludrocortisone.
* No coexisting medical conditions in the opinion of the investigator that would preclude participation in the study.

Exclusion Criteria:

* Current or history of active or chronic hepatitis, including symptomatic viral hepatitis A, B, or C.
* Any active infection.
* Evidence of active malignancy.
* Serious or uncontrolled co-existent non-malignant disease.
* Receiving systemic glucocorticoids for any reason other than for the treatment of 21-hydroxylase deficiency.
* Any disorders that require treatment with anticonvulsants.
* Patients of child-bearing potential who are not willing to use a method of birth control during the study and for 3 months after the end-of-study.
* Women who are pregnant or breast-feeding.
* Genotypes associated with non-classic congenital adrenal hyperplasia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The minimum dose of abiraterone acetate required to decrease serum androstenedione to the age-appropriate range for adult women with 21-hydroxylase deficiency | Up to Day 7 of each treatment period.
  Normalization or reduction of age-appropriate androstenedione levels will be determined by the mean of the androstenedione values measured on Study Days 6 and 7 of the treatment period.

SECONDARY OUTCOMES:
Mean serum concentrations of androstenedione | Up to Day 8 of each treatment period.
Mean serum concentrations of 17-hydroxyprogesterone | Up to Day 8 of each treatment period.
Mean plasma concentrations of renin activity | Up to Day 8 of each treatment period.
Mean serum concentrations of testosterone | Up to Day 8 of each treatment period.
Urine concentrations of androsterone | Up to Day 8 of each treatment period.
Urine concentrations of etiocholanolone | Up to Day 8 of each treatment period.
Maximum plasma concentration (Cmax) of abiraterone | Up to Day 8 of each treatment period.
Time to reach the maximum plasma concentration (tmax) of abiraterone | Up to Day 8 of each treatment period.
Area under the plasma concentration-time curve from time 0 to 24 hours postdose (AUC24) of abiraterone | Up to Day 8 of each treatment period.
Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration (AUClast) of abiraterone | Up to Day 8 of each treatment period.
Time to last quantifiable plasma concentration (Tlast) of abiraterone | Up to Day 8 of each treatment period.
Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of abiraterone | Up to Day 8 of each treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C., Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (3):
- United States (3):
  - Chicago, Illinois
  - Ann Arbor, Michigan
  - Dallas, Texas

REFERENCES:
- See also: An Open-Label, Multiple-Dose, Dose-Finding Study of Abiraterone Acetate in Adult Women With 21-Hydroxylase Deficiency — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2559&filename=CR100007_CSR.pdf